CLINICAL TRIAL: NCT05464602
Title: The Effect of Aromatherapy on Postoperative Pain, Sleep Quality and Physiological Parameters in Laparoscopic Cholecystectomy Patients
Brief Title: The Effect of Aromatherapy in Laparoscopic Cholecystectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Seda Akutay, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Erciyessbf
Record Dates: First submitted 2022-06-14; First posted 2022-07-19 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cholecystectomy; Aromatherapy
MeSH Terms: interventions — lavender oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group Lavender (Experimental): Each patient in this group received inhalation aromatherapy of lavender oil.
  Interventions: Other: Intervention group Lavender
- Intervention group Geranium (Experimental): Each patient in this group received inhalation aromatherapy of geranium oil.
  Interventions: Other: Intervention group Geranium
- Control group (No Intervention): Each patient in this group did not receive any additional treatment.

INTERVENTIONS:
Other: Intervention group Lavender — This group received inhalation aromatherapy 2 drops of lavender oil from aromastone for a total of 3 days, one day before the operation, the day of the operation and the first day after the operation.
  Other Names: Lavender oil
  Arms: Intervention group Lavender
Other: Intervention group Geranium — This group received inhalation aromatherapy 2 drops of geranium oil from aromastone for a total of 3 days, one day before the operation, the day of the operation and the first day after the operation.
  Other Names: Geranium oil
  Arms: Intervention group Geranium

SUMMARY:
Pain experienced before and after surgery in patients undergoing laparoscopic cholecystectomy adversely affects physiological parameters and sleep quality. This randomized controlled study was conducted to examine the effects of preoperative and postoperative inhalation lavender and geranium essential oil on patients undergoing laparoscopic cholecystectomy on pain, sleep, and physiological parameters. The study was completed with 3 groups and 150 people, namely the geranium oil group (n=50), lavender oil group (n=50) and control group (n=50). The ethics committee approval, informed consent of the individuals and the institutional permission were obtained. In the study, data were collected using the patient identification form, Richard-Campbell Sleep Scale and visual analog scale. Chi-square test,repeated measures one-way analysis of variance, and Spearman correlation analysis tests were used to assess the data. In the comparisons, the value of p<0.05 was accepted as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Hospitalized for laparoscopic cholecystectomy surgery,
* Alzheimer's, dementia etc. no disease,
* Having no perception problems (sense of smell, vision, hearing loss),
* Hospitalized the day before the operation,
* Patients who continue to stay in the hospital for at least one night after the operation will be included in the study.

Exclusion Criteria:

* Having any respiratory system disease (COPD, Asthma, etc.),
* Disturbed by the smell of essential oils,
* Any allergic diagnosis and history,
* Using anxiolytic, antidepressant,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | change from baseline score at the end of three day
  The range of 0 (zero) and 10cm is determined on a ruler. 0 (zero) means "no pain" and 10 means "worst possible pain". The patient is asked to mark the place that expresses the pain on the line. The distance marked by the patient is measured by taking the initial distance of zero.

SECONDARY OUTCOMES:
The Richards-Campbell Sleep Questionnaire | change from baseline score at the end of three day
  The Richard Campbell Sleep Questionnaire is a 6-item scale that evaluates the depth of sleep, the time to fall asleep, the frequency of awakening, the time to stay awake, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart with scores between 0 and 100. If the total mean score obtained from the scale is between "0-25", it indicates very bad sleep, between "26-75" indicates moderate sleep, and between "76-100" indicates very good sleep. The higher the score obtained from the scale, the higher the sleep quality of the patient is considered.

OTHER OUTCOMES:
Physiological parameter (Blood Pressure) | change from baseline score at the end of three day
  The systolic and diastolic blood pressures of the patients were recorded by the researchers the day before, the day of surgery, and the day after surgery.
Physiological parameter(Heart rate) | change from baseline score at the end of three day
  The heart rate of the patients was recorded by the researchers the day before the surgery, the day of the surgery, and the day after the surgery.
Physiological parameter(Respiratory rate) | change from baseline score at the end of three day
  The respiratory rate of the patients was recorded by the researchers the day before the surgery, the day of the surgery, and the day after the surgery.
Physiological parameter(SPO2) | change from baseline score at the end of three day
  The SPO2 of the patients was recorded by the researchers the day before the surgery, the day of the surgery, and the day after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan

REFERENCES:
- [Background] Saritas S, Kavak F, Savas B. The effect of lavender oil on anxiety levels of patients before laparoscopic cholecystectomy. Complement Ther Clin Pract. 2018 Aug;32:51-54. doi: 10.1016/j.ctcp.2018.05.003. Epub 2018 May 5. No abstract available. PMID 30057057
- [Background] Hwang E, Shin S. The effects of aromatherapy on sleep improvement: a systematic literature review and meta-analysis. J Altern Complement Med. 2015 Feb;21(2):61-8. doi: 10.1089/acm.2014.0113. Epub 2015 Jan 13. PMID 25584799
- [Background] Abdelhakim AM, Hussein AS, Doheim MF, Sayed AK. The effect of inhalation aromatherapy in patients undergoing cardiac surgery: A systematic review and meta-analysis of randomized controlled trials. Complement Ther Med. 2020 Jan;48:102256. doi: 10.1016/j.ctim.2019.102256. Epub 2019 Nov 23. PMID 31987220
- [Background] Lillehei AS, Halcon LL, Savik K, Reis R. Effect of Inhaled Lavender and Sleep Hygiene on Self-Reported Sleep Issues: A Randomized Controlled Trial. J Altern Complement Med. 2015 Jul;21(7):430-8. doi: 10.1089/acm.2014.0327. Epub 2015 Jun 2. PMID 26133206
- [Background] Bikmoradi A, Seifi Z, Poorolajal J, Araghchian M, Safiaryan R, Oshvandi K. Effect of inhalation aromatherapy with lavender essential oil on stress and vital signs in patients undergoing coronary artery bypass surgery: A single-blinded randomized clinical trial. Complement Ther Med. 2015 Jun;23(3):331-8. doi: 10.1016/j.ctim.2014.12.001. Epub 2014 Dec 11. PMID 26051567
- [Derived] Akutay S, Doner A, Ceyhan O, Baykan M, Saz A. Aromatherapy Improves Pain, Sleep and Physiological Parameters in Laparoscopic Cholecystectomy Patients: A Single-Blind, Parallel Group, and Randomized Controlled Trial. Chin J Integr Med. 2025 Jun 10. doi: 10.1007/s11655-025-3823-z. Online ahead of print. PMID 40490599